CLINICAL TRIAL: NCT03076853
Title: Medication Assessment Through Real Time Information eXchange - Distributed Pharmaceutical Record System
Acronym: MATRIX-DPRS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 13-PREPS-01
Record Dates: First submitted 2017-02-27; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Patients With Pharmaceutical Record

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Pharmaceutical Record
  Interventions: Other: Opening of the Pharmaceutical Record

INTERVENTIONS:
Other: Opening of the Pharmaceutical Record — After a first prescription without the pharmaceutical record, the study investigator has to open the pharmaceutical record to obtain some additional data. After, he has to choose between maintain or modify his first prescription.

SUMMARY:
The aim of MATRIX-DPRS is to assess the clinical and organizational impacts of the use of the medication record, opened, filled and managed by pharmacists (from private office and hospital units) by hospital physicians in private and public healthcare establishments (volunteers), for three clinical contexts: anaesthesiology visit before surgery, medications abuse and emergency hospitalization, medications and elderly hospitalisations.

DETAILED DESCRIPTION:
As part of the national 2012 PREPS call for proposals, a multidisciplinary research team was set up to design and develop methods in order to evaluate the efficiency and the performance of health data information systems. This team is composed of physicians and researchers in medical informatics, hospital information systems, biostatistics, process analysis and management in healthcare, ergonomics and usability. This study was aimed to evaluate the clinical and organizational impacts of the use of a new source of information brought by the pharmaceutical record, promoted by the national committee of pharmacists. This record is opened and filled for each patient by the pharmacist. It contains all the medication sold (prescribed by physician and OTC) by the patient. This record is used by almost all the private pharmacists. The French Health Ministry was looking for an evaluation of this new source of information by hospital physicians in order to be applied by any healthcare institution or organization wishing to evaluate the added value of its investments or recommendations (example: ARS (French Regional Health Agency), DGOS (French Directorate General of Health Services), etc.) in the information system.

ELIGIBILITY:
Inclusion Criteria:

Concerning Anesthesia department:

* Patients in pre-anesthesia consultation for scheduled intervention.

Concerning Emergencies department:

* Patients admitted for fainting fit

Regarding patients hospitalized in geriatrics:

* Patients admitted to geriatrics

Exclusion Criteria:

* Minors
* Patients without administrative or judicial freedom if the authorization of the legal representative can not be collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Anesthesia, Emergency and Geriatric departments with Pharmaceutical Record
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2016-04-03 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Modification of the medical prescription linked to the use of the pharmaceutical record | 3 months
  The primary outcome measure is to evaluate the impact of the use of the pharmaceutical record on th medical prescription. The doctor writes a first medical prescription without using the pharmaceutical record and a second with the pharmaceutical record.The changes are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No